CLINICAL TRIAL: NCT00884299
Title: Nutritional Enhancement in COPD: Randomized, Controlled Trial
Brief Title: Nutritional Enhancement in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: ARGALASTI HEALTH CENTRE (Unknown)
Responsible Party: LIANA KERANIS, ARGALASTI HEALTH CENTRE
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LK19021970DM
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Lung function; Chronic obstructive pulmonary disease; Antioxidants
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Free diet
- Diet rich in antioxidants (Experimental): Diet with increased consumption of foods containing antioxidants such as fresh fruits, fruit juices and vegetables. Patients in this arm will be seen regularly in the outpatient clinic where there will be informed for the potential beneficial effects of fruits and vegetables in health status by two members of the study team (attending physician and specialist nurse). At baseline and at each visit it is clearly explained to them that the dietary goal is to increase fresh fruit /fruit juices/vegetable consumption of at least one portion per day compared to baseline and to maintain this regime throughout the 3-year study period.
  Interventions: Dietary Supplement: Diet rich in antioxidants

INTERVENTIONS:
Dietary Supplement: Diet rich in antioxidants — Dietary intervention based on diet with increased consumption of foods containing antioxidants such as fresh fruits, fruit juices and vegetables. Patients are advised by a physician and a specialist nurse during regular scheduled outpatient clinic visits to increase fresh fruit /fruit juices/vegetable consumption of at least one portion per day compared to baseline and to maintain this regime throughout the study period.
  Arms: Diet rich in antioxidants

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by increased oxidative stress which aggravates airway and systemic inflammation. Previous studies suggested that dietary factors such as ample consumption of antioxidants might have beneficial effects in lung function in COPD patients.

The investigators' primary aim is therefore to investigate prospectively whether a nutritional intervention consisted of diet rich in antioxidants such as fresh fruits and vegetables, would significantly affect lung function decline in COPD patients compared to a free diet.

Methods: This is a 3-year prospective study, incorporating a run-in period of six months and outpatient clinic visits, scheduled every 6 months. Consecutive sampling was used to recruit 120 patients with COPD. At baseline and at each visit all patients were evaluated for respiratory symptoms, dietary habits, medication used and pulmonary function. Patients will be randomized either to a diet based on increased consumption of foods containing antioxidants (fresh fruits and vegetables), intervention group (IG) or, to a free diet, control group (CG).

The investigators hypothesize that the results from the study will suggest that a diet rich in antioxidants may be associated with improvement in lung function in COPD patients. In this respect dietary interventions should be considered in the management of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to the GOLD definition*
* Ability to perform spirometry.

(*Pauwels RA, Buist AS, Calverley PM, et al. Global strategy for the diagnosis, management and prevention of Chronic Obstructive Pulmonary disease. NHLBI/WHO Global initiative for Chronic Obstructive Lung Disease (GOLD). Workshop summary. Am J Respir Crit Care Med 2001; 163(5):1256-1276.)

Exclusion Criteria:

* A history of lung cancer, bronchial asthma or other respiratory disease
* Continuous use of systemic steroids more than 30 days prior was used as exclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Lung function decline | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: LIANA KERANIS, MD, Principal Investigator — University of Thessaly, Medical School
Locations (1):
- Argalasti Health Centre-University of Thessaly, Volos, Thessaly, Greece

REFERENCES:
- [Derived] Keranis E, Makris D, Rodopoulou P, Martinou H, Papamakarios G, Daniil Z, Zintzaras E, Gourgoulianis KI. Impact of dietary shift to higher-antioxidant foods in COPD: a randomised trial. Eur Respir J. 2010 Oct;36(4):774-80. doi: 10.1183/09031936.00113809. Epub 2010 Feb 11. PMID 20150206